CLINICAL TRIAL: NCT00931034
Title: The Effect of South Beach Diet™ Using South Beach Diet™ Products Compared to the American Diabetic Association Diabetes Meal Plan on Body Weight and Satiety in Overweight Diabetic Women
Brief Title: Effect of South Beach Diet (SBD™) Using SBD™ Products Compared to the American Diabetic Association (ADA) Diabetes Meal Plan on Body Weight and Satiety in Diabetic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Richard Black, PhD/VP, Nutrition, Kraft Foods
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07SWHK
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: South Beach Diet™; overweight; obesity; satiety; weight loss; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Weight Loss; Diabetes Mellitus | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- South Beach Diet with SBD Products (Active Comparator)
  Interventions: Behavioral: South Beach Diet with South Beach Diet Products
- ADA Diabetes meal plan (Active Comparator)
  Interventions: Behavioral: American Diabetes Association Diabetes Meal Plan

INTERVENTIONS:
Behavioral: South Beach Diet with South Beach Diet Products
  Arms: South Beach Diet with SBD Products
Behavioral: American Diabetes Association Diabetes Meal Plan
  Arms: ADA Diabetes meal plan

SUMMARY:
The purpose of this study is to examine the effectiveness of the South Beach Diet and products compared to the American Diabetic Association Diabetes Meal Plan.

ELIGIBILITY:
Inclusion Criteria:

1. Female age 18 to 55 years
2. Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result
3. Healthy as determined by laboratory results and medical history
4. Waist circumference > 87 cm
5. Stable weight defined as < 4.5 kg gained or lost in past year
6. Agreement to maintain current level of physical activity throughout the study
7. Diagnosed with Type II diabetes mellitus with fasting blood glucose 100 - 250 mg/dl (5.6 - 13.9 mmol/L)
8. Ability to comprehend and complete the questionnaires and forms
9. Agreement to comply with study procedures, test article consumption, and has access to a microwave oven
10. Voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Use of prescription or over the counter products known to effect weight including but not limited to the following:

   * megestrol acetate;
   * somatropin;
   * sibutramine;
   * orlistat;
   * paroxetine;
   * dextroamphetamine;
   * methylphenidate;
   * atomoxetine;
   * quetiapine;
   * olanzepine;
   * risperidone, within 4 weeks of randomization and during the trial
3. Unstable medication for diabetes mellitus (Dosage must be stable for 90 days prior to randomization), use of insulin is exclusionary
4. Alcohol use > 2 standard alcoholic drinks per day
5. Significant cardiac history defined as a history of:

   * myocardial infarction (MI);
   * coronary angioplasty or bypass graft(s);
   * valvular disease or repair;
   * unstable angina pectoris;
   * transient ischemic attack (TIA);
   * cerebrovascular accidents (CVA);
   * congestive heart failure; or
   * coronary artery disease (CAD)
6. History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission for more than 5 years are acceptable.
7. Uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
8. Unstable renal and/or liver disease
9. History of alcohol or drug abuse within the past year
10. Unstable psychiatric disorder requiring hospitalization within the past 6 months
11. Immunocompromised individuals such as subjects that have undergone organ transplantation or subjects diagnosed with human immunodeficiency virus (HIV)
12. History of hemoglobinopathies such as sickle cell anemia or thalassemia, sideroblastic anemia
13. Participation in another clinical research trial within 30 days prior to randomization and during the trial
14. Significant abnormal liver function as defined as AST and/or ALT > 2 x ULN, and/or bilirubin > 2 x ULN
15. Serum creatinine > 125 umol/L
16. Anemia of any etiology defined as hemoglobin < 110 g/L
17. Uncontrolled and/or untreated thyroid disorder
18. Unstable medications (Dosage must be stable for 90 days prior to randomization)
19. History of food allergies or sensitivities, including lactose intolerance
20. Vegetarians
21. Cognitively impaired and/or unable to give informed consent
22. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline to week 24 | 24 weeks

SECONDARY OUTCOMES:
Assess the satiety response to the individual diets | 24 weeks
Analyze circumference measurements & body composition; blood glucose, HbA1c, insulin, lipid profile, blood pressure & questionnaire responses on food cravings and quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Study Director — KGK Science Inc.
Locations (6):
- United States (6):
  - Medicus Research, Northridge, California
  - SIBR Research, Bradenton, Florida
  - Miami Research Associates, Miami, Florida
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - Rochester Clinical Research Inc, Rochester, New York
  - Chase Wellness & Research Center, Virginia Beach, Virginia